CLINICAL TRIAL: NCT06927869
Title: Effect of Pully System Exercise in Management of Spasticity in Cerebral Palsy Children: A Randomized Clinical Trial
Brief Title: Pully System Exercise Role in Management of Spasticity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Sara Yousef Abdel Elglil Yousef Elsebahy, lecturer of pediatric physical therapy, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-193
Record Dates: First submitted 2025-02-11; First posted 2025-04-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
Keywords: pully system; cerebral palsy; spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): the l group will receive a standard care program.
  Interventions: Other: designed physical therapy , pully system exercise
- study (Experimental): study group will received pulley system exercises
  Interventions: Other: designed physical therapy , pully system exercise

INTERVENTIONS:
Other: designed physical therapy , pully system exercise — Participants assigned to the intervention group will engage in a specially designed physical therapy program focusing on pulley system exercises. The program is scheduled to occur three times per week, which is frequent enough to potentially induce meaningful improvements while allowing adequate rest between sessions to prevent fatigue and overtraining

SUMMARY:
The goal of this clinical trial is to investigate the effect of pully system exercise in in management of spasticity in cerebral palsy children

Does pully system exercise has role in management of spasticity in cerebral palsy children ?

Participants will:

The participants assigned to the control group will receive a standard care program. This program is designed to provide basic supportive therapies without the specialized pulley system exercises

DETAILED DESCRIPTION:
there are two groups one group will receive traditional physical therapy programme another group will receive pully system exercise

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria
* The degree of spasticity is (1) according to Modified Ashwarth's scale
* They able to understand orders given to them.
* All children evaluated before and after the suggested period of the physical therapy program (3months).

Exclusion Criteria:

* - No fixed deformities.
* They have neither visual nor auditory problems.
* They have neither perceptual nor cognitive problems.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
gross motor function of children with cerebral palsy using GMFMS | 3 months
  evaluate change that occurs over time in the gross motor function of children with cerebral palsy
pediatric balance scale | 3 months
  A 14-item criterion-referenced measure that examines functional balance in the context of everyday tasks in the pediatric population.

SECONDARY OUTCOMES:
spasticity with EMG | 3 months
  In assessing muscle tone it is important to consider all the inputs and outputs affecting it, using biomechanical-EMG techniques for measuring active tone

OTHER OUTCOMES:
erobic capacity | 3 months
  6m walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Elsalam university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided